CLINICAL TRIAL: NCT02856672
Title: A Randomized Prospective Controlled Trial Comparing the Laryngeal Tube Suction Disposable and the Supreme Laryngeal Mask Airway: The Influence of Head and Neck Position on Oropharyngeal Seal Pressure
Brief Title: Trial Comparing the Laryngeal Tube Suction Disposable and the Supreme Laryngeal Mask Airway
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bnai Zion Medical Center (Other Government)
Collaborators: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Principal Investigator, LUIS.GAITINI, M.D., Bnai Zion Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: BnaiZionMC-16-LG-001
Record Dates: First submitted 2016-07-25; First posted 2016-08-05 (Estimated); Last update posted 2016-08-05 (Estimated); Status verified 2016-08

CONDITIONS: Adverse Anesthesia Outcome
Keywords: Laryngeal Tube Supreme Laryngeal Mask Airway Leak Pressure

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Supreme Laryngeal Mask Airway (Active Comparator): Supreme Laryngeal Mask Airway
  Interventions: Device: Supreme Laryngeal Mask Airway; Device: Laryngeal Tube Suction Disposable
- Laryngeal Tube Suction Disposable (Active Comparator): Laryngeal Tube Suction Disposable
  Interventions: Device: Supreme Laryngeal Mask Airway; Device: Laryngeal Tube Suction Disposable

INTERVENTIONS:
Device: Supreme Laryngeal Mask Airway — Supreme Laryngeal Mask Airway
Device: Laryngeal Tube Suction Disposable — Laryngeal Tube Suction Disposable

SUMMARY:
The investigators study compared the Laryngeal Tube Suction-Disposable with the Supreme Laryngeal Mask Airway, hypothesizing that the two devices would provide adequate oropharyngeal seal pressure in different head and neck positions and perform similarly during pressure controlled ventilation in neutral position, despite differences in their structural design.

DETAILED DESCRIPTION:
Laryngeal Tube Suction Disposable, LTS-D (VBM Medizintechnik GmbH , Sulz, Germany) and Supreme Laryngeal Mask Airway, SLMA (Intavent Orthofix, Maidenhead, UK) are second generation, single-use, supraglottic airway devices( SADs), with added gastric access, for use in spontaneously and mechanically ventilated patients undergoing general anesthesia.

The effectiveness of the LTS-D and the SLMA has been well established; however, the oropharyngeal seal pressure of both devices in different head/neck positions and the performance of these devices using positive pressure ventilation have not been evaluated. Changing the head/neck position can alter the sealing capabilities of the SAD.

To the investigators best knowledge there are no studies comparing the oropharyngeal seal pressure in different head and neck position when using these devices.

ELIGIBILITY:
Inclusion Criteria:

* Patients ASA I and II with normal airways, for minor elective surgical

Exclusion Criteria:

* Age <18 yr, weight <50 kg, or > 100 kg , a known difficult airway, active gastro esophageal reflux disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2009-01; Primary Completion 2010-01 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Primary outcome oropharyngeal seal pressures, in cm H2O | 5 min
  Oropharyngeal leak pressure was determined by closing the expiratory valve of the anesthesia breathing system and a fixed gas flow of the 3 liters minute. The airway pressure at which an equilibrium was reached was noted( maximun allowed 40 cm H2O)

SECONDARY OUTCOMES:
Fiberoptic position | 5 min
  Scoring system of the fiberoptic view: ranged from grade 4 (full view of arytenoids and glottis), 3 (arytenoids and glottis partly visible), 2 (view of arytenoids, glottis or epiglottis), and 1 (no part of larynx identifiable).

OTHER OUTCOMES:
Sore throat | 30 minutes after admission in Post Anesthetic Operative Unit ( PACU) and 24 hours postoperatively
  Sore throat was assessed subjetively by the patient using the 0-10 Numeric Pain Rating Scale

CONTACTS AND LOCATIONS:
Overall Officials: Luis A Gaitini, M.D., Principal Investigator — Bnai Zion Medical Center and Hospital Italiano de Buenos Aires

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Somri M, Vaida S, Garcia Fornari G, Mendoza GR, Charco-Mora P, Hawash N, Matter I, Swaid F, Gaitini L. A randomized prospective controlled trial comparing the laryngeal tube suction disposable and the supreme laryngeal mask airway: the influence of head and neck position on oropharyngeal seal pressure. BMC Anesthesiol. 2016 Oct 6;16(1):87. doi: 10.1186/s12871-016-0237-7. PMID 27716165